CLINICAL TRIAL: NCT05494502
Title: Impact of Erector Spinae Plane Block With Adjuvant Dexmedetomidine on Chronic Postsurgical Pain in Breast Cancer Patients: a Two-center Randomized Controlled Trial
Brief Title: Impact of Erector Spinae Plane Block on Chronic Postsurgical Pain in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-191
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Neoplasms; Mastectomy; Nerve Block; Dexmedetomidine; Pain, Postoperative; Chronic Pain; Prognosis
Keywords: Breast cancer; Mastectomy; Erector spinae plane block; Dexmedetomidine; Postoperative pain; Chronic postsurgical pain; Long-term prognosis
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Experimental): Prior to general anesthesia, ultrasound guided erector spinae plane block (ESPB; performed with 0.5% ropivacaine 35 ml with dexmedetomidine 1microgram/kg) is performed at T2 level (15 ml) and T4 level (20 ml).
  Interventions: Procedure: Erector spinae plane block
- Control group (Sham Comparator): General anesthesia alone.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Erector spinae plane block — Prior to general anesthesia, ultrasound guided erector spinae plane block (ESPB; performed with 0.5% ropivacaine 35 ml with dexmedetomidine 1 microgram/kg) is performed at T2 level (15 ml) and T4 level (20 ml).
  Arms: Erector spinae plane block group
Procedure: Control group — General anesthesia alone.
  Arms: Control group

SUMMARY:
Chronic postsurgical pain (CPSP) has an incidence of 46% in patients after breast cancer surgery, which seriously affects patients' physiological and psychological function, as well as quality of life. Acute pain is an independent risk factor for persistent pain after surgery. Erector spinae plane block (ESPB) provided excellent perioperative analgesia in patients undergoing breast surgery. Dexmedetomidine as an adjuvant of local anesthetics prolongs the duration of peripheral nerve block and decreases the requirements of postoperative analgesia. The investigators hypothesize that, for breast cancer patients undergoing mastectomy, ESPB (with a combination of 0.5% ropivacaine 35 ml and dexmedetomidine 1 microgram/kg) can reduce the occurrence of CPSP. The purpose of this randomized controlled trial is to investigate the impact of ESPB with adjuvant dexmedetomidine on the incidence of CPSP in breast cancer patients after mastectomy. We will also observe the impact of ESPB on long-term survival in these patients.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP), defined as pain persisting or recurring for longer than three months after surgery, has an incidence of 46% in patients after breast cancer surgery. It seriously affects patients' physiological and psychological function, as well as quality of life. Acute pain is an independent risk factor for persistent pain after surgery.

As a core technique in multimodal analgesia, peripheral nerve block plays an important role in controlling acute postoperative pain in breast cancer patients; it may also prevent the occurrence of CPSP. In our previous trial, use of paravertebral block reduced CPSP at six months after breast cancer surgery; the effect was more prominent in the subgroup of patients following mastectomy. But conclusions can not be achieved until now. Regional anesthesia is also supposed to produce favorable effects on long-term oncological outcomes, possibly by relieving surgery-related stress response and immunosuppression. But, again, available evidences are conflicting regarding regional block and long-term cancer outcomes.

The erector spinae plane block (ESPB) was first described by Forero in 2016 and provides excellent perioperative analgesia with minimal side effect in patients undergoing thoracic, breast, and spinal surgeries. As one of the interfacial plane block techniques, the ESPB targets dorsal and ventral rami of the spinal nerves from T2-T7; it may produce effect by diffusing into the paravertebral and intercostal spaces and spreading in both cephalic and caudal directions.

Dexmedetomidine is a highly selective α2-adrenoceptor agonist with sedative, analgesic and anti-anxiety properties. When used as an adjuvant to local anesthetics, dexmedetomidine prolongs the duration nerve block and decreased the requirement of postoperative analgesia.

The investigators hypothesize that, for breast cancer patients undergoing mastectomy, ESPB (with 0.5% ropivacaine 35 ml combined with dexmedetomidine 1 microgram/kg) can reduce the occurrence of CPSP. The purpose of this randomized controlled trial is to investigate the impact of ESPB with adjuvant dexmedetomidine on the incidence of CPSP in breast cancer patients after mastectomy. We will also observe the effect of ESPB on long-term prognosis in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or over, but less than 85 years;
2. Scheduled to undergo mastectomy for primary unilateral breast cancer.

Exclusion Criteria:

1. Previous breast cancer surgery with an incision of >2 cm;
2. Chronic opioid dependence or long-term intake of analgesic medicines (>3 months);
3. Any contraindication to erector spinae plane block, including intrathoracic infection, infection at the puncture site, cancer invasion of the puncture site, severe spinal deformity, history of spinal surgery, and severe coagulopathy;
4. Inability to communicate in the preoperative period because of profound dementia, deafness, language barriers, or end-stage disease;
5. History of malignant tumor in other organs, or a current combination of malignant tumor of other organs;
6. History of coronary heart disease (diagnosed coronary stenosis, previous myocardial infarction, previous percutaneous coronary intervention or coronary artery bypass grafting); preoperative hepatic or renal impairment (alanine transaminase and/or aspartate transaminase ≥2 times of upper limit of normal, or serum creatinine>133 µmol/L); history of peptic ulcer or hemorrhage; ASA classification IV or above;
7. Allergy to ropivacaine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1206 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic postsurgical pain (CPSP) at 6 months after surgery | At 6 months after surgery
  CPSP is defined as pain persisting for at least three months after surgery that was not present before surgery or that had different characteristics, and other possible causes of pain were excluded (e.g., cancer recurrence, infection).
Progression-free survival (long-term outcomes) | Up to 3 years after surgery
  Progression-free survival is defined as the time from randomization to disease progression (recurrence or metastasis) or death from any cause.

SECONDARY OUTCOMES:
Incidence of chronic postsurgical pain (CPSP) at 3 and 12 months after surgery | At 3 and 12 months after surgery
  CPSP is defined as pain persisting for at least three months after surgery that was not present before surgery or that had different characteristics, and other possible causes of pain were excluded (e.g., cancer recurrence, infection).
Incidence of neuropathic pain at 3, 6, and 12 months after surgery | At 3, 6 and 12 months after surgery
  Neuropathic pain is defined as a score at or above 0 on the Neuropathic Pain Questionnaire Short-form. The questionnaire contains three items, i.e., tingling pain, numbness, and increased pain due to touch. Each item is scored from 0 (no pain) to 100 (worst pain imaginable), and multiplied by a discriminant function coefficient (tingling: 0.017, numbness: 0.015, increased pain to touch: 0.011). The total sum of these is added to a constant value (-1.302) to yield a final score ranging from -1.302 to 2.998, with a cutoff of ≥0 suggesting neuropathic pain.
Overall survival (long-term outcome) | Up to 3 years after surgery
  Overall survival is defined as the time from randomization to death from any cause.
Event-free survival (long-term outcome) | Up to 3 years after surgery
  Event-free survival is defined as the time from randomization to tumor recurrence/metastasis, re-hospitalization for any reason, or death from any cause.
Quality of life (long-term outcome) | At 1 year, 2 years, and 3 years after surgery
  Quality of life is assessed with the breast cancer-specific Quality of Life Questionnaire (EORTC QLQ-BR53). It consists of EORTC-C30 [a 30-item questionnaire that provides assessments of functional dimensions (physical, role, cognitive, emotional, social, fatigue, pain, nausea/vomiting, a global health), the total score ranges from 0 to 100, with higher score indicating better function] and EORTC-BR23 [a 23-item questionnaire that provides assessments of symptom dimensions (systemic therapy side effects, arm symptoms, breast symptoms, body image, sexual functioning, sexual enjoyment, feeling of upset due to hair loss, and future perspective), the total score ranges from 0 to 100,with higher score indicating worse symptom].

OTHER OUTCOMES:
Pain intensity within the first 3 postoperative days | At 1 hour, 6 hours, 1 day, 2 days, and 3 days after surgery.
  Pain intensity is assessed with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain, both at rest and with movement.
Subjective sleep quality within the first 3 postoperative days | At 1 hour, 6 hours, 1 day, 2 days, and 3 days after surgery.
  Subjective sleep quality is assessed with the numeric rating scale, an 11-point scale where 0=the best sleep quality and 10=the worst sleep quality.
Patient-reported quality of recovery | At day 1 after surgery
  Patient-reported quality of recovery is assessed with the Quality of Recovery-15 scale (QoR-15 scale, a 15-item scale to assess the patients' postoperative recovery in physical comfort, emotional state, physical independence, psychological support and pain. For each item, the score ranges from 0 to 10. The total score ranges from 0 to 150, with higher score indicating better recovery).
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of postoperative complications within 30 days | Up to 30 days after surgery
  Postoperative complications are generally defined as newly occurred medical conditions that are deemed harmful and required therapeutic intervention within 30 days after surgery.
Incidence of anxiety at 30 days after surgery | At 30 days after surgery
  Anxiety is defined as a score of 8 or above on the anxiety subscale of the Hospital Anxiety and Depression Scale.
Incidence of depression at 30 days after surgery | At 30 days after surgery
  Depression is defined as a score of 8 or above on the depression subscale of the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, M.D., Ph.D., Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Wang L, Cohen JC, Devasenapathy N, Hong BY, Kheyson S, Lu D, Oparin Y, Kennedy SA, Romerosa B, Arora N, Kwon HY, Jackson K, Prasad M, Jayasekera D, Li A, Guarna G, Natalwalla S, Couban RJ, Reid S, Khan JS, McGillion M, Busse JW. Prevalence and intensity of persistent post-surgical pain following breast cancer surgery: a systematic review and meta-analysis of observational studies. Br J Anaesth. 2020 Sep;125(3):346-357. doi: 10.1016/j.bja.2020.04.088. Epub 2020 Jun 28. PMID 32611524
- [Background] Saporito A, Aguirre J, Borgeat A, Perren A, Anselmi L, Poggi R, Minotti B, Cafarotti S, La Regina D, Ceruti S. Persistent postdischarge pain and chronic postoperative pain after breast cancer surgery under general anesthesia and single-shot paravertebral block: incidence, characteristics and impact on quality of life and healthcare costs. J Pain Res. 2019 Apr 16;12:1193-1199. doi: 10.2147/JPR.S195702. eCollection 2019. PMID 31114301
- [Background] Kojic K, Clarke H. Important considerations with respect to reducing the transition from acute to persistent postoperative pain. Expert Opin Pharmacother. 2021 May;22(7):779-782. doi: 10.1080/14656566.2021.1892073. Epub 2021 Feb 26. No abstract available. PMID 33634743
- [Background] Rabbitts JA, Palermo TM, Lang EA. A Conceptual Model of Biopsychosocial Mechanisms of Transition from Acute to Chronic Postsurgical Pain in Children and Adolescents. J Pain Res. 2020 Nov 24;13:3071-3080. doi: 10.2147/JPR.S239320. eCollection 2020. PMID 33262642
- [Background] Lavand'homme P. The progression from acute to chronic pain. Curr Opin Anaesthesiol. 2011 Oct;24(5):545-50. doi: 10.1097/ACO.0b013e32834a4f74. PMID 21772141
- [Background] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545
- [Background] Saadawi M, Layera S, Aliste J, Bravo D, Leurcharusmee P, Tran Q. Erector spinae plane block: A narrative review with systematic analysis of the evidence pertaining to clinical indications and alternative truncal blocks. J Clin Anesth. 2021 Feb;68:110063. doi: 10.1016/j.jclinane.2020.110063. Epub 2020 Oct 5. PMID 33032124
- [Background] Zhang Y, Liu T, Zhou Y, Yu Y, Chen G. Analgesic efficacy and safety of erector spinae plane block in breast cancer surgery: a systematic review and meta-analysis. BMC Anesthesiol. 2021 Feb 20;21(1):59. doi: 10.1186/s12871-021-01277-x. PMID 33610172
- [Background] Li Y, Wang B, Zhang LL, He SF, Hu XW, Wong GT, Zhang Y. Dexmedetomidine Combined with General Anesthesia Provides Similar Intraoperative Stress Response Reduction When Compared with a Combined General and Epidural Anesthetic Technique. Anesth Analg. 2016 Apr;122(4):1202-10. doi: 10.1213/ANE.0000000000001165. PMID 26991622
- [Background] Desai N, Kirkham KR, Albrecht E. Local anaesthetic adjuncts for peripheral regional anaesthesia: a narrative review. Anaesthesia. 2021 Jan;76 Suppl 1:100-109. doi: 10.1111/anae.15245. PMID 33426668
- [Background] Vorobeichik L, Brull R, Abdallah FW. Evidence basis for using perineural dexmedetomidine to enhance the quality of brachial plexus nerve blocks: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2017 Feb;118(2):167-181. doi: 10.1093/bja/aew411. PMID 28100520
- [Background] Perez-Gonzalez O, Cuellar-Guzman LF, Soliz J, Cata JP. Impact of Regional Anesthesia on Recurrence, Metastasis, and Immune Response in Breast Cancer Surgery: A Systematic Review of the Literature. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):751-756. doi: 10.1097/AAP.0000000000000662. PMID 28953508
- [Background] Ramirez MF, Cata JP. Anesthesia Techniques and Long-Term Oncological Outcomes. Front Oncol. 2021 Dec 8;11:788918. doi: 10.3389/fonc.2021.788918. eCollection 2021. PMID 34956903
- [Background] Dockrell L, Buggy DJ. The role of regional anaesthesia in the emerging subspecialty of onco-anaesthesia: a state-of-the-art review. Anaesthesia. 2021 Jan;76 Suppl 1:148-159. doi: 10.1111/anae.15243. PMID 33426658
- [Background] Zhang J, Chang CL, Lu CY, Chen HM, Wu SY. Paravertebral block in regional anesthesia with propofol sedation reduces locoregional recurrence in patients with breast cancer receiving breast conservative surgery compared with volatile inhalational without propofol in general anesthesia. Biomed Pharmacother. 2021 Oct;142:111991. doi: 10.1016/j.biopha.2021.111991. Epub 2021 Aug 27. PMID 34449311